CLINICAL TRIAL: NCT02028221
Title: Phase II Study of Metformin for Reduction of Obesity-Associated Breast Cancer Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1300000596; 1R01CA172444-01A1 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer Prevention
Keywords: Breast cancer prevention; metformin; Breast cancer risk reduction
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1 tablet daily by mouth X 4 weeks, then 1 tablet twice daily by mouth for the remaining duration of the trial (12 months)
  Interventions: Drug: Placebo
- Metformin (Experimental): metformin 850 mg 1 tablet taken by mouth daily X 4 weeks, then metformin 850 mg 1 tablet taken twice daily for the remaining duration of he intervention period.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin 850 mg 1 tablet taken by mouth daily X 4 weeks, then metformin 850 mg 1 tablet taken twice daily for the duration of he intervention period.
  Other Names: Glucophage; Glumetza; Fortamet
  Arms: Metformin
Drug: Placebo — 1 tablet daily by mouth X 4 weeks, then 1 tablet twice daily by mouth for the remaining duration of the trial (12 months)
  Arms: Placebo

SUMMARY:
Overweight and obesity are well established risk factors for breast cancer that develop after menopause. The increased postmenopausal breast cancer risk in women who are overweight or obese is likely to be attributed to multiple metabolic disturbances. Metformin is a commonly used medication in diabetics to stabilize blood sugar. Association studies and laboratory studies have shown its potential to reduce the risk for development of cancer, including breast cancer. Recent pilot clinical studies in breast cancer patients suggest that metformin may only be effective in overweight or obese women with metabolic disturbances. We propose to conduct a clinical study of metformin in overweight or obese premenopausal women with metabolic disturbances. Study participants will be randomly assigned to receive metformin or placebo for 12 months. The study will evaluate whether metformin can result in favorable changes in risk features that have been associated with increased breast cancer risk. The risk features that will be examined in our study include breast density, certain proteins and hormones, products of body metabolism, and body weight and composition. The study should help determine the potential breast cancer preventive activity of metformin in a growing population at risk for multiple diseases.

DETAILED DESCRIPTION:
High adiposity is a major risk factor for a number of chronic diseases, including type 2 diabetes, cardiovascular diseases, and certain types of cancer, including postmenopausal breast cancer. The increased postmenopausal breast cancer risk in women with high adiposity is likely to be attributed to multiple metabolic disturbances including altered circulating sex steroid hormones, hyperinsulinemic insulin resistance, altered expression and secretion of adipokines from adipose tissue, increased production of pro-inflammatory cytokines, and increased oxidative stress.

Metformin, a widely used antidiabetic drug, exerts favorable effects on multiple metabolic disturbances which may lead to reduction of breast cancer risk in women with high adiposity. In addition, metformin may exert a direct effect in mammary tissue through the activation of the AMP-activated protein kinase signaling pathway, leading to an antiproliferative effect and induction of apoptosis. Recent case control and cohort studies found that treatment with metformin appears to substantially reduce the risk for development of cancer in diabetics, including breast cancer. There are a number of ongoing clinical trials of metformin in breast cancer patients. However, applicability of these trials to at risk healthy women requires further research and the concurrent or prior cancer treatments in these trials hinder the evaluation of metformin as a single agent for breast cancer risk reduction. In addition, recent clinical and animal studies suggest that metformin may only exert tumor suppressive effects in metabolic phenotypes of high adiposity and metabolic disturbances.

A Phase II randomized, double-blind, placebo-controlled trial of metformin in overweight/obese premenopausal women who have metabolic syndrome will be conducted. This study population is at increased risk for postmenopausal breast cancer and has a high prevalence of metabolic disturbances. The overall objective of this study is to determine its potential effects on reduction of obesity-associated breast cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* 21-54 years of age
* Have a BMI of 25 kg/m2 or greater
* No change in menstrual patterns for the past 6 months preceding the time of registration
* Waist circumference ≥ 35 inches or ≥ 31 inches for Asian Americans, individuals with polycystic ovary syndrome, or individuals with non-alcoholic fatty liver disease.
* Have at least one other component of metabolic syndrome (103) reported below:

  * Elevated triglycerides (≥ 150 mg/dL (1.7 mmol/L) or on drug treatment for elevated triglycerides
  * Reduced HDL-C (< 50 mg/dL (1.3 mmol/L) or on drug treatment for reduced HDL-C
  * Elevated blood pressure (≥ 130 Hg systolic blood pressure or ≥85 mm Hg diastolic blood pressure or on antihypertensive drug treatment in a patient with a history of hypertension
  * Elevated fasting glucose (≥100 mg/dL)
* Mammogram negative for breast cancer within the 12 months preceding the time of registration for women ≥ 50 years of age
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Postmenopausal women

  * Amenorrhea for at least 12 months (preceding the time of registration), or
  * History of hysterectomy and bilateral salpingo-oophorectomy, or
  * At least 55 years of age with prior hysterectomy with or without oophorectomy, or
  * Age 35 to 54 with a prior hysterectomy without oophorectomy OR with a status of ovaries unknown with documented follicle-stimulating hormone level demonstrating elevation in postmenopausal range
* Women who are pregnant, planning pregnancy within the next year, or breastfeeding
* On treatment with any drug for diabetes
* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any illness that would limit compliance with study requirements
* Have received chemotherapy and/or radiation for any malignancy (excluding non-melanoma skin cancer and cancers confined to organs with removal as only treatment) in the past 5 years (preceding the time of registration)
* Have received other investigational agents within the past 3 months (preceding the time of registration)
* Have a history of lactic acidosis or risk factors for lactic acidosis
* Have significant renal disease or dysfunction (creatinine ≥ 1.4 mg/dL)
* Have significant hepatic dysfunction (bilirubin ≥ 1.5 x ULN unless with Gilberts syndrome or AST/ALT ≥ 3 x ULN)
* Have a history of alcoholism or high alcohol consumption (average of > 3 standard drinks/day)
* Have a history of allergic reactions to metformin or similar drugs
* Have a history of severe claustrophobia
* Have electrically, magnetically, or mechanically activated implants including cardiac pacemaker, cochlear implants, magnetic surgical clips or prostheses
* Have breast implants

Ages: 21 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Chow, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Tapia E, Villa-Guillen DE, Chalasani P, Centuori S, Roe DJ, Guillen-Rodriguez J, Huang C, Galons JP, Thomson CA, Altbach M, Trujillo J, Pinto L, Martinez JA, Algotar AM, Chow HS. A randomized controlled trial of metformin in women with components of metabolic syndrome: intervention feasibility and effects on adiposity and breast density. Breast Cancer Res Treat. 2021 Nov;190(1):69-78. doi: 10.1007/s10549-021-06355-9. Epub 2021 Aug 12. PMID 34383179
- [Derived] Martinez JA, Chalasani P, Thomson CA, Roe D, Altbach M, Galons JP, Stopeck A, Thompson PA, Villa-Guillen DE, Chow HH. Phase II study of metformin for reduction of obesity-associated breast cancer risk: a randomized controlled trial protocol. BMC Cancer. 2016 Jul 19;16:500. doi: 10.1186/s12885-016-2551-3. PMID 27430256

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 75 | 76
Completed | 62 | 56
Not Completed | 13 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (8.6) | 39.9 (7.9) | 39.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 34 | 55
  Not Hispanic or Latino | 54 | 41 | 95
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 62 | 64 | 126
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 75 | 76 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change in Breast Density at 6 Months
Description: change of dense breast volume at 6 months
Time Frame: baseline, 6 months
Population: Analysis was performed on participants who provided baseline and 6 month breast density measures
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 41 | 38
cm^3 | -5.45 (48.91) | -13.71 (56.69)

2. Primary Outcome: Change in Breast Density at 12 Months
Description: Change in dense breast volume at 12 months
Time Frame: Baseline, 12 months
Population: Analysis was performed on participants who provided baseline and 12-month breast density measures
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 39
cm^3 | -12.11 (68.11) | -14.75 (47.84)

3. Secondary Outcome: Change From Baseline in Serum Insulin Levels at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: The number of participants analyzed refers to the number of participants with baseline data
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 74 | 76
uIU/ml
  Baseline | 14.6 (8.2) | 13.5 (8.7)
  6 months: number analyzed (Participants) | 63 | 60
  6 months | 14.0 (8.0) | 11.9 (8.0)
  12 months: number analyzed (Participants) | 62 | 56
  12 months | 13.1 (7.5) | 11.7 (8.1)

4. Secondary Outcome: Change From Baseline in Serum IGF-1 to IGFBP-3 Ratio at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: The number of participants analyzed refers to the number of participants with baseline data
Measure: Mean (Standard Deviation); unit: data presented as ratio; no unit
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 74 | 76
data presented as ratio; no unit
  Baseline | 0.178 (0.063) | 0.170 (0.061)
  6 months: number analyzed (Participants) | 63 | 60
  6 months | 0.178 (0.065) | 0.169 (0.061)
  12 months: number analyzed (Participants) | 62 | 56
  12 months | 0.171 (0.063) | 0.165 (0.060)

5. Secondary Outcome: Change From Baseline in Serum Testosterone Levels at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: Data were not collected
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Serum Leptin to Adiponectin Ratio at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: The number of participants analyzed refers to the number of participants with baseline data
Measure: Mean (Standard Deviation); unit: data presented as ratio; no unit
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 74 | 76
data presented as ratio; no unit
  Baseline | 0.023 (0.025) | 0.028 (0.051)
  6 months: number analyzed (Participants) | 63 | 60
  6 months | 0.022 (0.024) | 0.025 (0.047)
  12 months: number analyzed (Participants) | 62 | 56
  12 months | 0.021 (0.024) | 0.026 (0.052)

7. Secondary Outcome: Change From Baseline in Body Weight at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: The number of participants analyzed refers to the number of participants with baseline data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 75 | 76
kg
  Baseline | 102.3 (16.3) | 101.5 (18.9)
  6 months: number analyzed (Participants) | 63 | 60
  6 months | 102.1 (16.0) | 99.6 (19.2)
  12 months: number analyzed (Participants) | 62 | 56
  12 months | 103.2 (15.9) | 99.3 (19.4)

8. Secondary Outcome: Change From Baseline in Waist Circumference at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: The number of participants analyzed refers to the number of participants with baseline data
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 75 | 76
cm
  Baseline | 110.3 (11.4) | 111.2 (12.5)
  6 months: number analyzed (Participants) | 63 | 60
  6 months | 111.6 (11.3) | 108.9 (12.7)
  12 months: number analyzed (Participants) | 62 | 56
  12 months | 111.8 (10.9) | 108.3 (12.9)

9. Secondary Outcome: Change From Baseline in Serum IGF-2 Levels at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: Data were not collected
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Change From Baseline in Plasma Metabolomics Profile at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: Data were not collected
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Change From Baseline in Metabolomics Profile in Nipple Aspirate Fluid at 6 and 12 Months
Time Frame: baseline, 6 months, 12 months
Population: Data were not collected
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Metformin
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 7/75 | 1/76
Other Adverse Events (participants affected / at risk) | 61/75 | 67/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Metformin (N=76)
Renal colic (Renal and urinary disorders) | 0 | 1
Delusions (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine pain (Reproductive system and breast disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Metformin (N=76)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Bloating (Gastrointestinal disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 8 | 5
Diarrhea (Gastrointestinal disorders) | 15 | 28
Dyspepsia (Gastrointestinal disorders) | 11 | 14
Flatulence (Gastrointestinal disorders) | 9 | 2
Gastritis (Gastrointestinal disorders) | 4 | 2
Gastrointestinal disorders, other (Gastrointestinal disorders) | 8 | 8
Gastrointestinal pain (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 9 | 22
Stomach pain (Gastrointestinal disorders) | 4 | 9
Vomiting (Gastrointestinal disorders) | 8 | 3
Fatigue (General disorders) | 2 | 4
Flu like symptoms (General disorders) | 15 | 10
Bronchial infection (Infections and infestations) | 4 | 2
Otitis media (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 4 | 6
Upper respiratory infection (Infections and infestations) | 19 | 12
Urinary tract infection (Infections and infestations) | 6 | 4
Vaginal infection (Infections and infestations) | 4 | 0
Bruising (Injury, poisoning and procedural complications) | 5 | 2
Weight loss (Investigations) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 9
Headache (Nervous system disorders) | 13 | 16
Anxiety (Psychiatric disorders) | 4 | 2
Breast pain (Reproductive system and breast disorders) | 8 | 9
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Surgical and medical procedures, other (Surgical and medical procedures) | 4 | 4
Hypertension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02028221/Prot_SAP_000.pdf